CLINICAL TRIAL: NCT07169838
Title: Optimizing the Clinical Use of Perinatal Medical Waste: A Cost-Effectiveness Analysis of Fetal Stem Cell Production
Brief Title: Comparative Study of Perinatal Tissues for Clinical-Grade Mesenchymal Stem Cell Production and Cost-Effectiveness
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Copuroglu, M.D., Kayseri City Hospital
Other Study IDs: KayseriCityHospital; 28/2023 (Other: Eskişehir Osmangazi University Ethics Committee)
Record Dates: First submitted 2025-08-23; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Regenerative Medicine; Stem Cell Banking; Perinatal Medical Waste; Umbilical Cord Stem Cells
Keywords: Mesenchymal Stem Cells; Perinatal Medical Waste; Umbilical Cord; Stem Cell Banking; Cost-Effectiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women at term delivery providing perinatal tissue samples: Samples from this single cohort were divided into five tissue categories (amniotic fluid, amniotic membrane, umbilical cord, placental fragments, whole placenta) for comparative analysis of mesenchymal stem cell yield, sterility, and cost-effectiveness.
  Interventions: Other: Perinatal Tissue Collection

INTERVENTIONS:
Other: Perinatal Tissue Collection — Collection of perinatal medical waste (amniotic fluid, amniotic membrane, umbilical cord, placenta) at the time of term delivery for laboratory-based mesenchymal stem cell isolation and analysis. No therapeutic or interventional procedure was performed on participants.

SUMMARY:
This observational laboratory-based study was conducted to evaluate the clinical feasibility and cost-effectiveness of mesenchymal stem cell (MSC) production from perinatal medical waste, including umbilical cord, amniotic fluid, amniotic membrane, and placenta. A total of 160 tissue samples were collected from women delivering at term, and standardized protocols were applied for microbial sterility testing, MSC isolation, and cost analysis under Good Manufacturing Practice (GMP) conditions. The study compared MSC yield, contamination rates, and total processing costs across tissue types.

DETAILED DESCRIPTION:
Perinatal medical waste, including the umbilical cord, amniotic fluid, amniotic membrane, and placenta, represents a promising and ethically acceptable source of mesenchymal stem cells (MSCs). Unlike bone marrow or adipose-derived MSCs, which require invasive procedures and are limited by donor morbidity and age-related decline, perinatal tissues are collected non-invasively at the time of delivery and are usually discarded. This study was designed to optimize the clinical use of such tissues by systematically comparing their feasibility for large-scale MSC banking under Good Manufacturing Practice (GMP) conditions.

This prospective observational study was conducted between January and June 2023 at Eskişehir Osmangazi University and Kayseri City Hospital. A total of 160 perinatal tissue samples were collected at term deliveries, including amniotic fluid, amniotic membrane, umbilical cord (Wharton's jelly), whole placenta, and placental fragments. Samples were transferred to the GMP-compliant Cellular Therapy and Stem Cell Production Center for laboratory processing. Microbial contamination was assessed using the automated BACTEC™ FX system. MSCs were isolated through tissue-specific protocols, expanded in culture to passage 3, and characterized based on morphology and adherence criteria established by the International Society for Cellular Therapy (ISCT).

Quantitative outcomes included viable MSC yield per sample, sterility outcomes, and proliferative capacity. A detailed cost-effectiveness analysis was also performed, incorporating procurement, transportation, storage, reagents, disposables, and technician labor. Costs were standardized per 1×10⁶ viable MSCs and expressed in U.S. dollars according to the average 2023 exchange rate.

ELIGIBILITY:
Inclusion Criteria:

* Female participants only
* Age between 18 and 45 years
* Singleton, uncomplicated term pregnancies (≥37 weeks of gestation)
* Delivery by either elective cesarean section or spontaneous vaginal birth
* Written informed consent obtained prior to sample collection

Exclusion Criteria:

* Presence of maternal infection at the time of delivery
* Known fetal malformations or chromosomal abnormalities
* Placental abnormalities (e.g., previa, abruption)
* Preterm labor (<37 weeks)
* Any maternal comorbidity that may compromise tissue quality (e.g., uncontrolled diabetes, hypertension, autoimmune disease)
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants only, as the study involved collection of perinatal tissues (amniotic fluid, membranes, umbilical cord, placenta) at the time of childbirth.
Study Population: The study population consisted of 160 healthy women with uncomplicated singleton pregnancies who delivered at term (≥37 weeks) at Kayseri City Hospital and Eskişehir Osmangazi University Hospital in Türkiye. Participants were aged between 18 and 45 years. Perinatal tissues, including amniotic fluid, amniotic membrane, umbilical cord, and placenta, were collected immediately after delivery as medical waste, with no additional intervention applied. All participants provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Viable Mesenchymal Stem Cell Yield | Within 4 weeks after sample collection.
  The average number of viable mesenchymal stem cells (MSCs) isolated per perinatal tissue sample (×10⁶ cells per sample).

SECONDARY OUTCOMES:
Microbial Contamination Rate | Within 48 hours after collection.
  Proportion of perinatal tissue samples testing positive for microbial growth using the BACTEC™ FX system.
Cost per Million Viable MSCs | Calculated during the study period (January-June 2023).
  Average total cost (USD) of producing 1×10⁶ viable MSCs, including procurement, storage, isolation, and sterility testing.
Population Doubling Time (PDT) | Assessed at day 6-8 of culture expansion.
  The proliferative capacity of MSCs at passage 3, calculated as population doubling time (hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No